CLINICAL TRIAL: NCT04193748
Title: Evaluation of Topical Pomegranate Extracts in Management of Oral Lichen Planus (A Randomized Clinical Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Lecturer of Oral Medicine and Periodontology, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FacultyofDentistryCairoUni
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Oral Lichen Planus
Keywords: pomegranate, seeds, peel, topical, Oral lichen planus, pain, OHIP-14.
MeSH Terms: conditions — Lichen Planus, Oral; Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The clinical outcomes were assessed by an investigator masked about the treatment modality that has been used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): Topical triamcinolone acetonide 0.1% available commercially (Kenacort- in orabase) has been used. Topical corticosteroid treatment has be repeated four times per day for four weeks.
  Interventions: Drug: Topical pomegranate seeds and peel extracts
- Group S (Experimental): Topical pomegranate seeds extract treatment has been repeated four times per day for four weeks.
  Interventions: Drug: Topical pomegranate seeds and peel extracts
- Group P (Experimental): Topical pomegranate peel extract treatment has been repeated four times per day for four weeks.
  Interventions: Drug: Topical pomegranate seeds and peel extracts

INTERVENTIONS:
Drug: Topical pomegranate seeds and peel extracts — Topical pomegranate seeds and peel extracts in the form of gel

SUMMARY:
This study was conducted to estimate the hypothesis that the Pomegranate Extracts have no role in management of oral lichen planus

DETAILED DESCRIPTION:
Lichen planus is a common chronic mucocutaneous disease of uncertain origin that has been shown to affect 0.5% to 2.2% of various populations. The treatment options for OLP are numerous and include topical and systemic agents. Steroids were found effective in management of OLP with contraindicated use in some systemic diseases and with multiple side effects with its prolonged use. Pomegranates have been known for hundreds of years for their multiple health benefits, including anti-inflammatory activity. The recent surge indicates that pomegranates and their extracts may serve as natural alternatives to drugs which can offer a possible management of OLP decreasing pain and discomfort associated with this chronic condition.The aim of this study was the evaluation of the effect of topical pomegranate extracts in management of oral lichen planus lesions (OLP).

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion criteria were patients of both sexes with 18 to 60 years old in age with atrophic type OLP and signed the informed consent

Exclusion Criteria:

* Patients who excluded from the study were smokers, pregnant, lactating ladies and patients under topical and systemic steroids during the last two months. Uncontrolled diabetic patients or hypertension in addition to hepatic and cardiac patients were not included. In addition, any previous history of allergy to pomegranate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | 4 weeks
  Pain assessment scale

SECONDARY OUTCOMES:
Sign score | 4 weeks
  Score for clinical improvement of the signs
OHIP-14 questionnaire | 4 weeks
  evaluate the oral health related quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Oral Medicine and Periodontology Department, Cairo
  - Faculty of Dentistry, Cairo University, Giza

IPD SHARING:
Plan to Share IPD: No
Because the research not published yet.